CLINICAL TRIAL: NCT02779660
Title: Effect of Remote Ischemic Preconditioning on Electrophysiological and Biomolecular Parameters in Non-valvular Paroxysmal Atrial Fibrillation: RIPPAF Study
Acronym: RIPPAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jedrzej Kosiuk (Other)
Responsible Party: Sponsor-Investigator, Jedrzej Kosiuk, MD Jedrzej Kosiuk, Heart Center Leipzig - University Hospital
Organization: Heart Center Leipzig - University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RIPPAF V1
Record Dates: First submitted 2016-05-12; First posted 2016-05-20 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIPC-Group (Experimental): After randomization patients will undergo 3 sessions of RIPC (Remote ischemic preconditioning) intervention: I) on preoperative day, II) 1 h before and III) directly before the blood sample collection and invasive measurement of electrophysiological parameters.
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- Control-Group (Placebo Comparator): After randomization patients will undergo 3 sessions of sham-intervention: I) on preoperative day, II) 1 h before and III) directly before the blood sample collection and invasive measurement of electrophysiological parameters.
  Interventions: Procedure: sham-intervention

INTERVENTIONS:
Procedure: Remote ischemic preconditioning (RIPC) — RIPC will be induced by the application of 3 short episodes (5 minutes) of forearm ischemia by cuff sphygmomanometer inflation separated by 5 minutes of reperfusion.
  Arms: RIPC-Group
Procedure: sham-intervention — In the control group the cuff will be inflated for 3 times at 10 mm Hg for 5 minutes with 5-minute intervals
  Arms: Control-Group

SUMMARY:
The aim of the study is to examine the effect of RIPC on physiological parameters in non-valvular paroxysmal atrial fibrillation. Furthermore the study will provide a unique bio-date base for further analysis of molecular and genetic mechanisms responsible for observed results.

The potential effect of RIPC on AF inducibility and/or prothrombotic activity might be implemented as additional treatment component to reduce AF burden and minimize thromboembolic risk.

Interim Analysis will be done after 73 patients.

ELIGIBILITY:
Inclusion Criteria:

* planned invasive Atrial Fibrillation ablation

Exclusion Criteria:

* AF in ECG at Admission
* history of AF ablation
* age <18
* pregnancy
* neoplastic disorders
* acute or systemic inflammation, autoimmune diseases
* documented atrial flutter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
inducibility of Atrial Fibrillation by high-rate pacing of 20 s | during the Atrial Fibrillation Ablation procedure
sustainability of Atrial Fibrillation measured in seconds | during the Atrial Fibrillation Ablation procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Herzzentrum Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kosiuk J, Langenhan K, Stegmann C, Uhe T, Dagres N, Dinov B, Kircher S, Richter S, Sommer P, Bertagnolli L, Bollmann A, Hindricks G. Effect of remote ischemic preconditioning on electrophysiological parameters in nonvalvular paroxysmal atrial fibrillation: The RIPPAF Randomized Clinical Trial. Heart Rhythm. 2020 Jan;17(1):3-9. doi: 10.1016/j.hrthm.2019.07.026. Epub 2019 Jul 26. PMID 31356986